CLINICAL TRIAL: NCT07013734
Title: Patient Positioning and Its Influence on BIS, NOL, and Cerebral Oxygenation in Anesthetized Patients
Status: Not yet recruiting | Type: Observational
Sponsor: Ciusss de L'Est de l'Île de Montréal (Other)
Responsible Party: Sponsor
Other Study IDs: 2025-3803
Record Dates: First submitted 2025-04-30; First posted 2025-06-10 (Actual); Last update posted 2025-06-10 (Actual); Status verified 2025-04

CONDITIONS: Monitoring of Depth of Anesthesia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this observational study is to find out how changes in body position during surgery might affect brain monitoring results in patients who are under general anesthesia.The main question it aims to answer is:

- Does patient positioning have an impact on Bispectral Index (BIS) and Nociception Level (NOL) index monitoring (which are values of awareness in anesthesized patients).

Participants will undergo their surgery as planned, except for these extra features:

* Extra monitors placed to check brain activity, pain response, and brain oxygen levels.
* Before the surgery, while the patient is asleep, the patient's table will be moved into two different positions for 2 minutes each to see if the values on the monitor change.

Participants will then have to answer a short questionnaire after surgery about their memories before and after the anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* Fully consented, adult patients above 18 years old;
* Supine positioning during the surgery;
* Surgery requiring patient positioning with Vacuform mats.

Exclusion Criteria:

* Patient with Body Mass Index (BMI) ≥ 35;
* Patients over 80 years old.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients from Maisonneuve-Rosemont Hospital undergoing elective surgery.
Sampling Method: Probability Sample
Enrollment: 64 (Estimated)
Dates: Start 2025-08 (Estimated); Primary Completion 2026-03 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Variation in Bispectral Index (BIS) | Perioperative period

SECONDARY OUTCOMES:
Variation of Nociception Level (NOL) Index | Perioperative period
Variation of the patient's cerebral saturation measured with cerebral oximetry | Perioperative period